CLINICAL TRIAL: NCT00720135
Title: A Phase I Study of De-Immunized DI-Leu16-IL2 Immunocytokine in Patients With B-Cell Non-Hodgkin Lymphoma
Brief Title: Fusion Protein Cytokine Therapy After Rituximab in Treating Patients With B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03131; NCI-2010-01228; CDR0000598679 (Registry Identifier: PDQ); P50CA107399 (NIH)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Anaplastic Large Cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — Rituximab; Flow Cytometry; Immunohistochemistry; Enzyme-Linked Immunosorbent Assay; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive DI-Leu16-IL2 immunocytokine IV over 4 hours on 4 consecutive Wednesdays. Patients with detectable CD20-positive B-cells pretreatment also receive rituximab IV on 4 consecutive Tuesdays. Treatment repeats every 6-8 weeks for up to a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: DI-Leu16-IL2 immunocytokine; Biological: rituximab; Other: flow cytometry; Other: immunohistochemistry staining method; Other: pharmacological study; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay; Genetic: reverse transcriptase-polymerase chain reaction

INTERVENTIONS:
Biological: DI-Leu16-IL2 immunocytokine — Given IV
  Other Names: de-immunized anti-CD20-IL-2 immunocytokine DI-Leu16-IL-2; DI-Leu16-IL-2
Biological: rituximab — Given IV
  Other Names: C2B8 Monoclonal Antibody; IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: flow cytometry — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR

SUMMARY:
RATIONALE: Biological therapies, such as fusion protein cytokine therapy, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving fusion protein cytokine therapy together with rituximab may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of fusion protein cytokine therapy when given after rituximab in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of DI-Leu16-IL2 (DI-Leu16-IL2 immunocytokine) following peripheral blood B cell depletion with rituximab in patients with B-cell NHL.

II. To investigate the optimal biological dose (OBD) of DI-Leu16-IL2 following peripheral blood B cell depletion with rituximab in patients with B-cell NHL, which may differ from the MTD.

III. To describe the toxicities associated with the proposed DI-Leu16-IL2 regimen.

SECONDARY OBJECTIVES:

I. To evaluate the immunogenicity as measured by the induction of DI-Leu16-IL2-specific antibodies.

II. To evaluate the pharmacokinetics of DI-Leu16-IL2. III. To document any clinical responses associated with the proposed therapy and survival endpoints of the enrolled patients.

OUTLINE: This is a dose-escalation study of DI-Leu16-IL2 immunocytokine.

Patients receive DI-Leu16-IL2 immunocytokine IV over 4 hours on 4 consecutive Wednesdays.

Patients with detectable CD20-positive B-cells pretreatment also receive rituximab IV on 4 consecutive Tuesdays.

Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion

* Patients with CD20-expressing B cell NHL that is relapsed or refractory to standard therapy; CLL/SLL with peripheral blood leukemia/lymphoma cells and high-grade lymphomas (i.e., lymphoblastic lymphoma/Burkitt lymphoma) are excluded
* Patients must have received prior Rituxan
* Measurable disease; in the absence of lymphadenopathy, splenomegaly with defects or measurable extramedullary disease is acceptable; however, bone marrow involvement alone will not be included in the study
* Age >=18 years and <=65 physiologic years of age
* KPS >= 70%
* Life expectancy >= 12 weeks
* Serum creatinine =< 1.5 mg/dl
* Total WBC >= 3000/ul or absolute neutrophil count (ANC) >= 1000/ul
* Lymphocyte count >= 0.2 x 10^3/ul
* Platelet count >= 75,000/ul
* Hematocrit >= 25% or hemoglobin >= 9 g/100 ml
* Alanine aminotransferase (ALT) =< 2.5 x UNL
* Aspartate aminotransferase (AST) =< 2.5 x UNL
* Total bilirubin (TBili) < 1.5 x UNL
* Sodium, potassium, and phosphorus within normal limits
* Chest x ray (CXR) within 4 weeks prior to Day 1 with no evidence of pulmonary congestion, pleural effusions, pulmonary fibrosis, or significant emphysema; if results are questionable, subjects would have additional lung function testing to exclude clinically relevant restriction or obstruction; subjects must have an FEV-1 and DLCO of at least 65% and 50% of expected, respectively
* Electrocardiogram (12-lead ECG)
* Echocardiogram (or MUGA) with normal left ventricular function
* Cardiac stress test (e.g., stress thallium scan, stress echocardiography) with normal results if subject is suspected to have coronary artery disease
* Fasting blood glucose (FBG) < 160 and hemoglobin (Hgb) A1C < 7% for subjects with diabetes mellitus (DM) or borderline DM
* Women of procreative potential must have negative pregnancy test within the 2-week screening phase prior to Cycle 1, and all subjects of procreative potential must use adequate birth control throughout the study; subjects of procreative potential are defined as any fertile male, and any female who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy or bilateral oophorectomy) or is not post-menopausal, defined as age-related amenorrhea >= 12 months
* Provide written informed consent prior to any screening procedures

Exclusion

* Evidence of CNS lymphoma or lymphomatous meningitis
* Prior treatment with IL-2
* Type I hypersensitivity or anaphylactic reactions to murine proteins or to previous infusion of rituximab
* Pregnant or lactating female
* An immediate need for palliative radiotherapy or systemic corticosteroid therapy
* Known intercurrent infections (including hepatitis C virus [HCV] and HIV or other conditions), or clinical evidence of these conditions
* Actively infected with or chronic carriers of hepatitis B virus (HBV) as demonstrated by positive hepatitis B core antibody (HbcHb) or hepatitis B surface antigen (HbsAg); (subjects who are sero-positive only, i.e., surface antibody positive [HbsAg], are permitted)
* Other significant active infection
* Major surgery, chemotherapy, investigational agent, or radiation within 30 days of Day 1
* Uncontrolled hypertension (diastolic >= 100 mmHg) or hypotension (systolic =< 90 mmHg)
* History of repeated and clinically relevant episodes of syncope or other paroxysmal, ventricular, or other significant arrhythmias
* On ECG: a marked baseline prolongation of QT/QTc interval (> grade 2 QTc interval > 470 milliseconds)
* History of medically significant ascites requiring repetitive paracentesis
* Previous diagnosis of Addison's disease
* Previous diagnosis of autoimmune disease (exceptions: subjects with autoimmune thyroiditis or vitiligo may be enrolled)
* Organ transplant recipient
* History of prior therapy or a serious, uncontrolled medical disorder that in the investigator's opinion would impair participation in the study
* Known hypersensitivity to Tween-80 or human immunoglobulin
* Legal incapacity or limited legal capacity
* Patients with bulky lymph nodes (>= 10cm) or marked splenomegaly (i.e., extending into pelvis or crossing the midline)
* Positive anti-DI-Leu16-IL2 antibody assay (where positive is defined as > 10% of the radiolabeled DI-Leu16-IL2 reactive with the subject's serum)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of DI-Leu16-IL2 | 6 weeks post cycle 1 of treatment
Optimal biologic dose of DI-Leu16-IL2 | 6 weeks after final cycle of treatment
Toxicities associated with the DI-Leu16-IL2 regimen | 6 weeks after final cycle of treatment

SECONDARY OUTCOMES:
Immunogenicity as a result of DI-Leu16-IL2 administration | Within 2 weeks following a 4 week treatment period
Pharmacokinetics of DI-Leu16-IL2 administration | 6 weeks after final cycle of treatment
Clinical responses and survival | Within two weeks following completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States